CLINICAL TRIAL: NCT02756884
Title: Phase I/Phase II Safety and Preliminary Efficacy Study Using Low Frequency Ultrasound in Addition to Adipose Derived Stem Cells (ADSCs) in Patients With Moderate to Severe Lower Extremity Peripheral Arterial Disease (PAD)
Brief Title: Safety and Preliminary Efficacy of Adipose Derived Stem Cells and Low Frequency Ultrasound in PAD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arkansas Heart Hospital (Other)
Collaborators: SonaCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHH-2015-10
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LoFU and aADSC (Experimental): Low Frequency Ultrasound LFUS will be delivered in a non-sterile manner using a custom modified LFUS combined imaging/therapy probe. Adipose derived stem cells from the patient will be harvested through lipoaspiration. This solution will be injected intra-venous, intra-adventitia and intramuscular in the affected vessel and area after the administration of the low frequency ultrasound
  Interventions: Biological: LoFU and aADSC
- Adipose Derived Stem Cells (Active Comparator): Adipose derived stem cells from the patient will be harvested through lipoaspiration. This solution will be injected intra-venous, intra-adventitia and intramuscular in the affected vessel and area without the administration of the low frequency ultrasound
  Interventions: Biological: adipose derived stem cells

INTERVENTIONS:
Biological: LoFU and aADSC — Administration of low frequency ultrasound prior to administration of autologous adipose derived stem cells.
  Arms: LoFU and aADSC
Biological: adipose derived stem cells — control arm will only received the adipose derived stem cells.
  Arms: Adipose Derived Stem Cells

SUMMARY:
This is a single center, open label, prospective, randomized, controlled study in patients with non- revascularizable moderate or severe lower extremity Peripheral Arterial Disease (PAD) receiving autologous stem cells therapy (minimally manipulated). This study will enroll a maximum of 10 subjects in this study. The patients will be divided into two groups. One group will receive Adipose Derived Stem Cells (ADSCs) alone and the other group will receive low frequency ultrasound before the addition of ADSCs. The randomization will be 1:1. If the results of this pilot study are not clearly different, there will be a need for a phase II study to support the results.

Baseline, 6 week, 3 month and 6 month assessments of 6 min walking distance (6MWT), Ankle Brachial Indexes (ABIs)/Toe Brachial Indexes (TBIs), Transcutaneous Partial Oxygenation (TcPO2) and Rutherford assessments will be performed for the study group. Prior to the stem cell treatment, the ultrasound group patient will receive noninvasive transcutaneous pulsed focused ultrasound around the involved vessel(s) in the affected extremity. All patients will then receive 200 million autologous stromal vascular fraction cells containing adipose derived stem cell therapy: 1/3 of the cells will be delivered intra-venous proximal to the lesion (not retrograde), 1/3 of the cells will be delivered intra- adventitia proximal to the lesion and 1/3 of the cells will be delivered by intra- muscular injection along the vessel path (20-30 injections each separated by1.5 inch). Standard therapy for PAD patients will not be interrupted for the duration of the study. Standard therapy for PAD is defined as cardiovascular general measures like lifestyle changes, smoke cessation, exercise, cardiovascular rehabilitation, etc. All participants have already received maximal non-surgical therapy. Safety will be monitored on an ongoing basis.

DETAILED DESCRIPTION:
This is a single center, open label, prospective, randomized, controlled study in patients with non- revascularizable moderate or severe lower extremity PAD receiving autologous stem cells therapy. We will enroll a maximum of 10 subjects in this study. The patients will be divided into two groups. One group will receive ADSCs alone and the other group will receive low frequency ultrasound before the addition of ADSCs. The randomization will be 1:1. If the results of this pilot study are not clearly different, there will be a need for a phase II study to support the results.

Baseline, 6 week, 3 month and 6 month assessments of 6 min walking distance, ABIs/TBIs, TcPO2, Rutherford assessments will be performed for the study group. Prior to the stem cell treatment, the ultrasound group patient will receive noninvasive transcutaneous pulsed focused ultrasound around the involved vessel(s) in the affected extremity. All patients will then receive 100 to 200 million autologous adipose derived stem cell therapy: 1/3 of the cells will be delivered intra-venous proximal to the lesion (not retrograde), 1/3 of the cells will be delivered intra- adventitia proximal to the lesion and 1/3 of the cells will be delivered by intra- muscular injection along the vessel path (20-30 injections each separated by 1.5 inch). Standard therapy for PAD patients will not be interrupted for the duration of the study. Standard therapy for PAD is defined as cardiovascular general measures like lifestyle changes, smoke cessation, exercise, cardiovascular rehabilitation, etc. All participants have already received maximal non-surgical therapy. Safety will be monitored on an ongoing basis.

SUBJECT PARTICIPATION A screening evaluation to determine if a potential subject is suitable for participation in this trial will be conducted prior to enrollment and treatment by the Investigator. This includes obtaining written informed consent, collection of a complete medical history, including current and past medications, physical examination and clinical laboratory tests, PAD related testing (ABI/TBI, 6MWT, TcPO2, QoL questionnaires, etc.).

Eligible subjects will be randomized and treated at the Sponsor hospital as approved by the sponsor. Study medical staff will evaluate the patients upon admission according to the scheduled medical assessments to ensure eligibility of the subjects. Ultrasound group will receive LFUS over the affected limb (see page XIV). Intra-venous, intra-adventitia and intramuscular dosing of the autologous ADSC will occur on the morning of Day 0. Conscious sedation (I.V.) may be used during the tissue harvesting and intra-adventitia administration of the cells.. Subjects must remain in the clinic/hospital until they are clinically stable for discharge; subjects that are clinically stable will be discharged into the care of a responsible individual. Follow-up visits will occur at 6 weeks and 3 and 6 months post-treatment, and may occur with the patient's personal physician who will be provided the follow-up assessment forms. If this occurs, the Investigator and/or Sponsor or sponsor's designee may also contact the patient by telephone to collect follow-up safety information. Adverse events, concomitant medications, vital signs, clinical laboratory test results and physical examinations will be collected or conducted at follow-up visits according to the schedule of assessments (Appendix B). All previous medical care, including medications and rehabilitation, for the patient's current medical conditions will be continued as prescribed by the patient's personal physician(s). Use of other investigational agents or treatments is not allowed during this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females ≥18 years
2. Patients with a Rutherford classification of 3 or 4.
3. Non revascularizable lesions by balloon or stent angioplasty of the lower extremity SFA (Superficial femoral artery), Popliteal, AT (anterior tibial), PT (posterior tibial) or peroneal arteries. Non-revascularizable lesions will be determined based on a CT angiogram and/ or angiography.
4. Life expectancy greater than 6 months.
5. Ability to understand and provide signed informed consent.
6. Reasonable expectation that patient will receive standard post-treatment care and attend all scheduled safety follow-up visits
7. Written informed consent

Exclusion Criteria:

1. Immunosuppressive agents, including but not limited to, corticosteroids and steroidal anti- inflammatory agents (SAIDS)
2. Non-steroidal anti- inflammatory agents (NSAIDS)
3. Patients taking currently P2Y12 inhibitors or calcium channel blockers.
4. Uncontrolled seizure disorder
5. Dementia
6. Evidence or presence of immune deficiency.
7. Presence of any other clinically-significant medical condition, psychiatric condition, or laboratory abnormality that in the judgment of the Investigator or Sponsor would pose a safety risk to the subject
8. Participation in another study with an investigational drug or device within one month prior to treatment
9. Females known to be pregnant, lactating or having a positive pregnancy test (will be tested during screening) or planning to become pregnant during the study
10. Inability to comply with the conditions of the protocol.
11. Allergy to sodium citrate or any "caine" type of local anesthetic

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Safety measured by incidence of adverse events | 6 months
  The primary outcome will be the safety/tolerability of treatment with aADSC in patients with PAD as determined by the incidence and severity of adverse events and serious adverse events.

SECONDARY OUTCOMES:
Efficacy of stem cells in improving ABI | 6 months
  Changes in ABI reported as an entire number with two decimals (e.g. 1.00) from baseline
Efficacy of stem cells in improving 6MWT | 6 months
  Improvement in six minute walk test (6MWT) in meters when compared to baseline.
Efficacy of stem cells in improving the TcPO2 | 6 months
  improvement in Transcutaneous oxygen pressure (TcPO2) in mmHg as compared to baseline
Efficacy of stem cells in improving Quality of Life using EQ-5D 5L questionnaire | 6 months
  Improvement in overall quality of life as measured using the EQ-5D 5L questionnaire as compared to baseline.
Efficacy of stem cells in improving Quality of Life using the VascuQol questionnaire | 6 months
  Improvement in overall quality of life as measured using the VascuQol questionnaire as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Wong, MD, Principal Investigator — Arkansas Heart Hospital
Locations (2):
- United States (2):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Arkansas Site Management Services LLC, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tebebi PA, Burks SR, Kim SJ, Williams RA, Nguyen BA, Venkatesh P, Frenkel V, Frank JA. Cyclooxygenase-2 or tumor necrosis factor-alpha inhibitors attenuate the mechanotransductive effects of pulsed focused ultrasound to suppress mesenchymal stromal cell homing to healthy and dystrophic muscle. Stem Cells. 2015 Apr;33(4):1173-86. doi: 10.1002/stem.1927. PMID 25534849